CLINICAL TRIAL: NCT05245188
Title: Evaluation of Cognitive Performance in 4 Dairy Beverages
Acronym: COG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: UCAMCFE-00024
Record Dates: First submitted 2022-01-23; First posted 2022-02-17 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-01

CONDITIONS: Cognitive Performance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental Product 1 (Experimental): Consumption of 200 ml of product 1. Subjects will take this amount only on the day of the visit that they are to consume this product.
  Interventions: Other: Chocolate milk shakes - Product 1
- Experimental Product 2 (Experimental): Consumption of 200 ml of product 2. Subjects will take this amount only on the day of the visit that they are to consume this product.
  Interventions: Other: Chocolate milk shakes - Product 2
- Experimental Product 3 (Experimental): Consumption of 200 ml of product 3. Subjects will take this amount only on the day of the visit that they are to consume this product.
  Interventions: Other: Chocolate milk shakes - Product 3
- Experimental Product 4 (Experimental): Consumption of 200 ml of product 4. Subjects will take this amount only on the day of the visit that they are to consume this product.
  Interventions: Other: Chocolate milk shakes - Product 4

INTERVENTIONS:
Other: Chocolate milk shakes - Product 1 — 11.3 glucose
  Arms: Experimental Product 1
Other: Chocolate milk shakes - Product 2 — 8.84 glucose
  Arms: Experimental Product 2
Other: Chocolate milk shakes - Product 3 — 4.24 glucose
  Arms: Experimental Product 3
Other: Chocolate milk shakes - Product 4 — 4.36 glucose
  Arms: Experimental Product 4

SUMMARY:
The objective of the study is to evaluate the cognitive performance of 4 chocolate milk drinks.

DETAILED DESCRIPTION:
Subjects will make a total of 4 visits. Four visits in which they will drink a chocolate milkshake at each visit.

At each visit the subjects will have to come fasting, and they will have to perform the cognitive test at the time when they have their peak glycemic level.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes (10 men and 10 women).
* Subjects aged between 20 and 35 years.
* Subjects with a body mass index between 20 and 25 kg/m2.

Exclusion Criteria:

* Subjects suffering from diabetes mellitus or any chronic disease.
* Subjects with medical problems or a diagnosed psychiatric disorder.
* Subjects with alcohol abuse or excessive alcohol consumption (>3 glasses of wine or beer/day).
* Subjects consuming any pharmacological medication that may affect memory.
* Participation in another clinical trial in the three months prior to the study.
* Unwillingness or inability to comply with clinical trial procedures.
* Subjects whose condition does not make them eligible for the study according to the investigator's criteria.
* Pregnant or lactating women.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Cognitive performance | The test was carried out half an hour after consumption of the product, except for product 4, which was carried out 15 minutes after consumption.
  COMPASS cognitive test panel

SECONDARY OUTCOMES:
Depression, Anxiety and Stress | The test was carried out half an hour after consumption of the product, except for product 4, which was carried out 15 minutes after consumption.
  DASS21 test
Sleep quality | The test was carried out half an hour after consumption of the product, except for product 4, which was carried out 15 minutes after consumption.
  Pittsburgh test

CONTACTS AND LOCATIONS:
Overall Officials: Fco Javier López Román, Principal Investigator — Catholic University of Murcia
Locations (1):
- Catholic University of Murcia, Murcia, Spain